CLINICAL TRIAL: NCT01088477
Title: Imaging of ER Density to Guide and Improve Tailored Therapy for Acquired Anti-hormonal Resistant Breast Cancer
Status: Completed | Type: Observational
Sponsor: University Medical Center Groningen (Other)
Collaborators: Dutch Cancer Society (Other)
Responsible Party: Sponsor
Other Study IDs: RUG 2009-4529
Record Dates: First submitted 2010-03-16; First posted 2010-03-17 (Estimated); Last update posted 2024-05-06 (Actual); Status verified 2024-05

CONDITIONS: Breast Cancer
Keywords: Acquired anti-hormonal resistant breast cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Breast cancer patients with acquired anti-hormonal resistance
  Interventions: Other: Diagnostic intervention: Positron Emission Tomography with 16-alpha-[18-fluoro]-17betaestradiol

INTERVENTIONS:
Other: Diagnostic intervention: Positron Emission Tomography with 16-alpha-[18-fluoro]-17betaestradiol — In patients with acquired antihormonal resistance, eligible for estrogen therapy, a FES-PET scan will be made to determine FES-PET tumor uptake (which corresponds to estrogen receptor expression levels). Immediately after the FES-PET scan, all patients will start with a standard accepted dose of 2mg estradiol TID. Therapy response will be monitored by regular follow-up. RECIST criteria and clinical benefit will be used as criteria. In case of disease progression before end of the study period, estradiol treatment will be stopped.

SUMMARY:
In 50 breast cancer patients, heavily pretreated with anti-hormonal therapy, the investigators will evaluate the use of 16-alpha[18-fluoro]-17beta-estradiol positron emission tomography (FES-PET)as predictive biomarker for response to estrogen therapy.

DETAILED DESCRIPTION:
The estrogen receptor (ER) is expressed in approximately 70% of the breast carcinomas. In general, for these patients anti-hormonal therapy is the therapy of first choice. Despite good responses in 50-60% of the patients, unfortunately all patients develop (acquired) resistance. Patients with acquired anti-hormonal resistance can be subdivided into three different groups: (1) patients that have lost ER-expression (~25%), (2) patients with preserved ER-expression (~55%) and (3) patients with enhanced ER-expression (~30%). Several studies suggest different treatment strategies for these three different ER-phenotypes in antihormonal resistant breast cancer. In patients with acquired anti-hormonal resistance, ~30% of the patients still respond to hormone-additive therapy with estrogens. In vitro studies have shown estrogen-induced apoptosis in long-treated estrogen deprived cells (simulating aromatase inhibitor resistance). It is suggested that this estrogen-hypersensitivity is accompanied by increased ER-expression.

Whole-body imaging of ER-density is now possible with positron emission tomography with the 16-alpha[18-fluoro]-17beta-estradiol tracer (FES-PET). FES-PET has shown to be a predictive biomarker for response to first line anti-hormonal therapy.

In this study we will include 50 patients, heavily pretreated with anti-hormonal therapy. All patients will undergo FES-PET at baseline and start estrogen therapy. Investigators and patients will be blinded for FES-PET results. Responders and non-responders will be defined using RECIST criteria and clinical follow-up. After response has been determined, FES-PET results will be analyzed. We hypothesize that patients responding to estrogen therapy can be identified on basis of high ER-expression determined by FES-PET.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with the diagnosis of acquired anti-hormonal resistant advanced breast cancer showing progression after two or more lines of antihormonal treatment;
2. Treatment with estradiol will be started;
3. Age> 18 years;
4. ECOG performance status 0-2.

Exclusion Criteria:

1. Life Expectancy <3 months;
2. Uncontrolled CNS metastases;
3. History of thrombosis;
4. Uncontrolled hypercalcemia;
5. Treatment with any investigational drug within 30 days before start of study;
6. Serious uncontrolled concurrent illness, e.g. autoimmune disorders;
7. New York Hearth Association (NYHA) class III/IV congestive heart failure;
8. Dyspnea at rest due to any cause;
9. Pregnant or lactating women. Documentation of a negative pregnancy test must be available for pre-menopausal women with intact reproductive organs and for women less than two years after menopause;
10. Women of childbearing potential unless a) surgically sterile or b) using adequate measures of contraception.
11. Diabetes Mellitus

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Breast cancer patients with acquired anti-hormonal resistance, treated with at least 2 lines of anti-hormonal therapy
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2010-02; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Quantifying FES-uptake to predict response to estrogen therapy | 2 years
  FES-uptake (prior to estrogen therapy) of tumour lesions will be recorded for all patients.
  Patients will be prospectively categorized into responders and non-responders during standard follow-up (consisting of monthly visits, 3-monthly CT, and other techniques when indicated). Patients with complete response, partial response or stable disease for >6 months are defined as 'responders'.
  With ROC analysis we will determine the optimal cut-off value for FES-uptake to predict response to estrogen therapy.

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands

REFERENCES:
- [Background] Dehdashti F, Mortimer JE, Trinkaus K, Naughton MJ, Ellis M, Katzenellenbogen JA, Welch MJ, Siegel BA. PET-based estradiol challenge as a predictive biomarker of response to endocrine therapy in women with estrogen-receptor-positive breast cancer. Breast Cancer Res Treat. 2009 Feb;113(3):509-17. doi: 10.1007/s10549-008-9953-0. Epub 2008 Mar 9. PMID 18327670
- [Background] Ellis MJ, Gao F, Dehdashti F, Jeffe DB, Marcom PK, Carey LA, Dickler MN, Silverman P, Fleming GF, Kommareddy A, Jamalabadi-Majidi S, Crowder R, Siegel BA. Lower-dose vs high-dose oral estradiol therapy of hormone receptor-positive, aromatase inhibitor-resistant advanced breast cancer: a phase 2 randomized study. JAMA. 2009 Aug 19;302(7):774-80. doi: 10.1001/jama.2009.1204. PMID 19690310
- [Background] Linden HM, Stekhova SA, Link JM, Gralow JR, Livingston RB, Ellis GK, Petra PH, Peterson LM, Schubert EK, Dunnwald LK, Krohn KA, Mankoff DA. Quantitative fluoroestradiol positron emission tomography imaging predicts response to endocrine treatment in breast cancer. J Clin Oncol. 2006 Jun 20;24(18):2793-9. doi: 10.1200/JCO.2005.04.3810. Epub 2006 May 8. PMID 16682724